CLINICAL TRIAL: NCT04375462
Title: AspireAssist for Palliative Venting Gastrostomy in Malignant Bowel Obstruction Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left CCF
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE12219
Record Dates: First submitted 2020-03-24; First posted 2020-05-05 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Malignant Small Bowel Obstruction; Malignant Gastric Outlet Obstruction
MeSH Terms: interventions — Surveys and Questionnaires; goblet cell silencer inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AspireAssist (Experimental): Gastrostomy tubes will be placed 1-2 days after enrollment. Questionnaires will be completed at 7 and 30 days, and the AspireAssist group will have a clinic visit at 7 days to have the skin-port placed.
  All participants will be placed on a diet consisting of liquids and soft foods to prevent clogging of the gastrostomy tube
  Interventions: Device: AspireAssist device; Other: gastric outlet obstruction scoring system (GOOSS) questionnaire; Other: Modified Gastroparesis Cardinal Symptom Index (GCSI) questionnaire; Other: Patient satisfaction and ease of use survey
- Standard PEG (Active Comparator): Gastrostomy tubes will be placed 1-2 days after enrollment. Questionnaires will be completed at 7 and 30 days All participants will be placed on a diet consisting of liquids and soft foods to prevent clogging of the gastrostomy tube
  Interventions: Device: Standard decompressive PEG tube; Other: gastric outlet obstruction scoring system (GOOSS) questionnaire; Other: Modified Gastroparesis Cardinal Symptom Index (GCSI) questionnaire; Other: Patient satisfaction and ease of use survey

INTERVENTIONS:
Device: AspireAssist device — Allows for aspiration of gastric contents into a receptacle or the toilet to prevent symptoms of nausea, vomiting, and to prevent aspiration.
  Device is placed endoscopically in an identical fashion to a standard PEG tube G 1-2 days after enrollment
  Arms: AspireAssist
Device: Standard decompressive PEG tube — Allows for gastric drainage to prevent symptoms of nausea, vomiting, and to prevent aspiration.
  Device is placed endoscopically 1-2 days after enrollment
  Arms: Standard PEG
Other: gastric outlet obstruction scoring system (GOOSS) questionnaire — Gastric outlet obstruction scoring system (GOOSS) questionnaire
  Both groups will receive the questionnaires via a phone call
Other: Modified Gastroparesis Cardinal Symptom Index (GCSI) questionnaire — Modified Gastroparesis Cardinal Symptom Index (GCSI) questionnaire
  Both groups will receive the questionnaires via a phone call
Other: Patient satisfaction and ease of use survey — Patient satisfaction and ease of use survey
  Both groups will receive the questionnaires via a phone call

SUMMARY:
Individuals with cancer causing an intestinal or stomach obstruction often require gastric drainage to prevent symptoms of nausea, vomiting, and to prevent aspiration. This is often achieved by a nasogastric (NG) tube, although prolonged NG tube use can lead to unwanted side effects like ulcers, bleeding, and they are generally uncomfortable. Gastric drainage through the use of a percutaneously placed endoscopic gastrostomy (PEG) tube has been used in people with cancer since the 1980s. This allows relief of symptoms of malignant bowel obstruction though venting of stomach contents. Decompressive PEG tubes are routinely used in individuals with malignant obstruction, although these tubes tend to get clogged from food blocking the tube.

The AspireAssist is a weight loss device that allows participants to remove a large amount of the food in their stomachs after each meal to help them to lose weight via an aspiration device attached to the abdominal portion of the tube which allows instillation of water into the stomach, followed by aspiration of the gastric contents into a receptacle or the toilet. The device is placed endoscopically in an identical fashion to a standard PEG tube. Although most commonly used for weight loss, the device is FDA cleared to be used as a venting tube as well.

The purpose of this study is to determine if the AspireAssist provides an improved quality of life when compared with a standard venting gastrostomy tube for participants with malignant bowel obstructions.

DETAILED DESCRIPTION:
This multicentered study will enroll participants into two cohorts of (study and control groups). The study group will undergo AspireAssist gastrostomy tube placement and the control group will undergo standard decompressive percutaneous gastrostomy tube placement. Individuals who present for venting gastrostomy placement in clinic or as consults will be approached for inclusion. Gastrostomy tubes will be placed 1-2 days after enrollment to allow for thoroughly consideration of inclusion by potential participants. Gastrostomy tube placement will be completed endoscopically in the standard "pull" method in both the AspireAssist and PEG groups. Questionnaires will be completed at 7 and 30 days.

The primary objective of this study is to evaluate to compare healthcare utilization, including major and minor tube related complications between the two groups. Secondary objectives of this study are to compare changes in the ability to eat and drink after placement of the gastrostomy tube and to evaluate changes in quality of life before and after gastrostomy tube placement.

ELIGIBILITY:
Inclusion Criteria:

* Malignant (cancer of any type) gastric or small bowel obstruction referred to surgery for placement of a venting gastrostomy tube for gastric decompression
* Able to demonstrate the ability to use the AspireAssist prior to placement

Exclusion Criteria:

* Those who are immobile and unable to at least sit up in bed to vent the gastrostomy tube.
* Undergoing placement of a gastrostomy tube for any other indication other than malignant small bowel or gastric outlet obstruction.
* Absolute contraindications to gastrostomy tube placement, such as occluding oral or esophageal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of tube related complications per day | at 30 days
  Number of tube related complications per day, including tube clogging, skin infection, dislodgement, etc.
Patient satisfaction and ease of use survey scores | At baseline
  Patient satisfaction and ease of use survey, with scores ranging from 0-15 with lower scores corresponding to higher satisfaction with the tube
Patient satisfaction and ease of use survey scores | At 7 days from the date of tube placement
  Patient satisfaction and ease of use survey, with scores ranging from 0-15 with lower scores corresponding to higher satisfaction with the tube
Patient satisfaction and ease of use survey scores | At 30 days from the date of tube placement
  Patient satisfaction and ease of use survey, with scores ranging from 0-15 with lower scores corresponding to higher satisfaction with the tube
Quality of life as measured by Edmonton Symptom Assessment System (ESAS) | At baseline
  Quality of life as measured by Edmonton Symptom Assessment System (ESAS), with scores ranging from 0-100 with higher scores corresponding to worse outcomes
Quality of life as measured by Edmonton Symptom Assessment System (ESAS) | At 7 days from the date of tube placement
  Quality of life as measured by ESAS, with scores ranging from 0-100 with higher scores corresponding to worse outcomes
Quality of life as measured by Edmonton Symptom Assessment System (ESAS) | At 30 days from the date of tube placement
  Quality of life as measured by ESAS, with scores ranging from 0-100 with higher scores corresponding to worse outcomes

SECONDARY OUTCOMES:
Number of decompressions per day | at 30 days
  Number of decompressions per day
Number of ED visits or readmissions for tube related problems | at 30 days
  Number of ED visits or readmissions for tube related problems
Number of calls or office visits for nausea or tube related issues | at 30 days
  Number of calls or office visits for nausea or tube related issues
Ability to eat/drink assessed via GOOSS | At baseline
  Ability to eat/drink assessed via GOOSS, with scores ranging from o to 3, with higher scores indicating higher levels of oral intake.
  Pre and postoperative GOOSS scores will be compared using Wilcoxon signed rank test with a p <0.05 being considered significant
Ability to eat/drink assessed via GOOSS | At 1 week from the date of tube placement
  Ability to eat/drink assessed via GOOSS, with scores ranging from o to 3, with higher scores indicating higher levels of oral intake.
  Pre and postoperative GOOSS scores will be compared using Wilcoxon signed rank test with a p <0.05 being considered significant
Ability to eat/drink assessed via GOOSS | At 30 days from the date of tube placement
  Ability to eat/drink assessed via GOOSS, with scores ranging from o to 3, with higher scores indicating higher levels of oral intake.
  Pre and postoperative GOOSS scores will be compared using Wilcoxon signed rank test with a p <0.05 being considered significant

CONTACTS AND LOCATIONS:
Overall Officials: Alisan Fathalizadeh, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study of 40 participants and IPD will not be shared